CLINICAL TRIAL: NCT05011747
Title: Long Term Surgical Outcomes of Viscotrabeculotomy in Pediatric Glaucoma Following Cataract Surgery
Brief Title: Viscotrabeculotomy in Pediatric Glaucoma Following Cataract Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Amr Mohammed Elsayed Abdelkader, Associate professor of ophthalmology, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Viscotrabeculotomy in GFCS
Record Dates: First submitted 2021-08-06; First posted 2021-08-18 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Glaucoma Congenital
Keywords: Pediatric glaucoma,; Trabeculotomy; Congenital cataract surgery
MeSH Terms: conditions — Hydrophthalmos

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- single-site VT group (Active Comparator): Viscotrabeculotomy is performed through a superonasal triangular scleral flap.
  Interventions: Procedure: single-site rigid probe viscotrabeculotomy (VT)
- two-site VT group (Active Comparator): Viscotrabeculotomy is performed through a superonasal and an inferotemporal triangular scleral flap.
  Interventions: Procedure: two-site rigid probe viscotrabeculotomy (VT)

INTERVENTIONS:
Procedure: single-site rigid probe viscotrabeculotomy (VT) — single-site VT by the rigid probe trabeculotome is performed through a superonasal triangular scleral flap.
  Arms: single-site VT group
Procedure: two-site rigid probe viscotrabeculotomy (VT) — Two-site VT by the rigid probe trabeculotome is performed through a superonasal and an inferotemporal triangular scleral flap.
  Arms: two-site VT group

SUMMARY:
Long term Surgical Outcomes of Viscotrabeculotomy in Pediatric Glaucoma Following Cataract Surgery.

Purpose:

This study aims to compare outcomes of single-site rigid probe viscotrabeculotomy (VT) to two-site VT in pediatric secondary glaucoma following cataract surgery.

Methods:

This is a comparative study was performed on patients aged ≤ 12 years and required surgery for glaucoma following congenital cataract surgery (GFCS) with or without intraocular lens (IOL) implantation. Eyes in which the trabeculotomy involves <180° of Schlemm's canal ,eyes that have synechial angle closure over ≥ 90° and eyes that have previous procedures other than lensectomy or IOL implantation are excluded from the study. Eyes are then randomized to undergo single-site VT or two-site VT using a random table. The two-site VT by the rigid probe trabeculotome is performed through a superonasal and an inferotemporal triangular scleral flap. Intraocular pressure (IOP), anti-glaucoma medications, complications and success rates at dates of follow up are all reported. Success is defined as IOP between 6-20 mmHg or 35% IOP reduction with or without topical anti-glaucoma medications and without visually-devastating complications or additional glaucoma surgery.

DETAILED DESCRIPTION:
Long term Surgical Outcomes of Viscotrabeculotomy in Pediatric Glaucoma Following Cataract Surgery.

Introduction:

Despite advances in congenital cataract management, secondary glaucoma (SG) remains a major postoperative sight-threatening complication, with open-angle glaucoma being the predominant type in both aphakic and pseudophakic children . Although the pathogenesis of glaucoma after cataract surgery remains unclear, several risk factors have been identified. These include early surgery, chronic postoperative inflammation , primary posterior capsulotomy , persistence of fetal vasculature , and microphthalmia .

However, the pathogenesis of the classic, open-angle type of glaucoma that develops on average 1.3-12.2 years following uneventful cataract surgery is still obscure. Mechanical collapse of the trabecular meshwork due to the loss of ciliary body tension could be one of the possible reasons. Some speculate that obstruction of the trabecular meshwork by inflammatory cells, lens remnants and vitreous-derived factors may result in delayed elevation in IOP. Arrest of postnatal angle maturation secondary to the surgical intervention could be a contributing factor, especially that aphakic glaucoma is more likely to occur in patients who had lensectomy at a younger age, usually the first year of life. The incidence of secondary pediatric glaucoma after cataract surgery is not yet precisely identified. It ranges from 3%-41% depending on the follow-up period and the criteria chosen to define glaucoma . Management of paediatric glaucoma following cataract surgery (GFCS) is challenging. Trabeculectomy has a poor success rate and precludes the use of contact lenses, especially in the presence of thin, avascular, cystic blebs . Glaucoma drainage devices have a higher chance of success than trabeculectomy, but aphakic eyes have relatively higher rates of complications, especially suprachoroidal haemorrhage, if hypotony occurs particularly if buphthalmic. GDD-implanted eyes also carry a life-long risk of developing keratopathy secondary to endothelial decompensation from the tube end .Cyclodestructive procedures provide a temporizing treatment with occasional longterm control after multiple treatments. Yet, it is difficult to titrate with marked inflammation and a risk of phthisis, especially in microphthalmic eyes. Furthermore, it may be associated with chronic hypotony and may prejudice future surgery to failure. Angle surgery was first described as a surgical option in GFCS by Chen et al., yielding promising results in terms of IOP lowering and surgical success. Unlike bleb-based procedures, angle surgery addresses the more physiological outflow pathway through the trabecular meshwork and Schlemm's canal. Hence the risk of bleb-based complications such as infection, bleb leak, overfiltration and bleb dysthesia is reduced. With the growing evidence that circumferential trabeculotomy yields superior results to conventional 180° angle surgery in primary congenital glaucoma16, Freedman et al. retrospectively reported the results of microcatheter-assisted circumferential trabeculotomy in GFCS, achieving a 72% success rate. several reports in treatment of pediatric glaucoma have concluded that the use of viscoelastic materials during trabeculotomy may increase the success rate of the procedure by preventing ocular decompression, postoperative hemorrhage, anterior chamber shallowness, and adhesion of the incision lips or fibroblastic proliferation18.The purpose of the present study was to compare outcomes of single-site rigid probe viscotrabeculotomy (VT) Versus two-site VT in pediatric secondary glaucoma following cataract surgery.

Patients and methods:

This is a comparative study , performed on patients aged ≤ 12 years and required surgery for glaucoma following congenital cataract surgery (GFCS) with or without intraocular lens (IOL) implantation. The study will be conducted at the outpatient clinic of Mansoura Ophthalmic Center of Mansoura University in Mansoura, Egypt.

Eyes in which the trabeculotomy involves <180° of Schlemm's canal ,eyes that have synechial angle closure over ≥ 90° and eyes that have previous procedures other than lensectomy or IOL implantation are excluded from the study. Eyes are then randomized to undergo single-site VT or two-site VT using a random table. The two-site VT by the rigid probe trabeculotome is performed through a superonasal and an inferotemporal triangular scleral flap. The primary outcome of this study is compare the success rate in lowering IOP between the 2 surgical options; the single-site VT versus two-site VT. Success is defined as IOP between 6-20 mmHg or 35% IOP reduction with or without topical anti-glaucoma medications and without visually-devastating complications or additional glaucoma surgery.

The secondary clinical outcomes will include Intraocular pressure (IOP) control values, horizontal corneal diameter, axial length, cup- disc ratio, antiglaucoma medication, refractive error and postoperative complications in these 2 surgical procedures. Data will be analysed.

Statistical analysis:

All statistical analysis was accomplished using IBM SPSS version 20. Assessment of the data normality was done using both Histogram plot and Shapiro-Wilk's test. Wilcoxon test was used to compare the preoperative and postoperative variables in each group. The comparison between the two groups was done using Mann-Whitney test for numerical variables and Chi-square test for categorical variables. Kaplan-Meier survival curve was plotted to estimate the mean survival time and probabilities of failure at different follow-up stages in the both groups. For all tests, P value of less than 0.05 was considered significant.

ELIGIBILITY:
Inclusion Criteria:

-Patients aged ≤ 12 years and required surgery for glaucoma following congenital cataract surgery (GFCS) with or without intraocular lens (IOL) implantation.

Exclusion Criteria:

* Eyes in which the trabeculotomy involves <180° of Schlemm's canal.
* Eyes that have synechial angle closure over ≥ 90°.
* Eyes that have previous procedures other than lensectomy or IOL implantation.

Ages: 2 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
the success rate in lowering IOP | 3 years
  Success is defined as IOP between 6-20 mmHg or 35% IOP reduction with or without topical anti-glaucoma medications and without visually-devastating complications or additional glaucoma surgery.
  IOP was evaluted during each Follow up visit using applanation tonometry.

SECONDARY OUTCOMES:
Intraocular pressure (IOP) control values | 3 years
  measured at each follow up visit using tonopen ,icare or applantion tonometery
antiglaucoma medications. | 3 years
  The total number of antiglaucoma medications needed to control the IOP
postoperative complications | 3 years
  Include: Hyphaema with its grades, IOP spikes and Hypotony and possible inflammation or infections
horizontal corneal diameter. | 3 years
  Measured manually during follow visits using a caliber
axial length. | 3 yeras
  Measured by A scan mode of the US
cup- disc ratio. | 3 years
  Detected clinically and documented by fundus photo

IPD SHARING:
Plan to Share IPD: Yes
IPD will be provided as a supplementary digital content
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 3 years
Access Criteria: IPD will be provided as a supplementary digital content with publication